CLINICAL TRIAL: NCT06942143
Title: An Open-label, Phase I Clinical Trial of Autologous T Cells Transduced With NY-ESO-1 Antigen-specific High-affinity T Cell Receptors in NY-ESO-1-positive Patients With Advanced Solid Tumors
Brief Title: An Open-label, Phase I Clinical Trial of Super1 TCR-T in NY-ESO-1-positive Patients With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Guangzhou FineImmune Biotechnology Co., LTD. (Industry)
Collaborators: Sun Yat-sen University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FIT002-IIT
Record Dates: First submitted 2025-03-25; First posted 2025-04-24 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-04

CONDITIONS: Sarcoma; Lung Cancers; Melanoma
Keywords: Cell therapy; Immunotherapy; Solid tumor; NY-ESO-1 TCR-T
MeSH Terms: conditions — Sarcoma; Lung Neoplasms; Melanoma

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Dose escalation was performed in a 3+3 design (Experimental): The Super1 TCR-T dose toxicity test was escalated according to the following dose (positive cells) escalation schedule:
  Level 1 Level 2 Level 3
  Interventions: Biological: Super1 TCR-T

INTERVENTIONS:
Biological: Super1 TCR-T — All participators received lymphoid-depleted preconditioning before Super1 TCR-T cells infusion. Super1 TCR-T cells were infused 3 days later. Concomitant administration of interleukin for 7 consecutive days.
  Other Names: NY-ESO-1 TCR-T

SUMMARY:
This study was a phase I safety and tolerability clinical trial conducted in a single-center, open-label, 3+3 design with dose escalation.

DETAILED DESCRIPTION:
After the subjects signed the informed consent form, the HLA genotype of the subjects was detected. After the HLA genotype was confirmed as A*02, the tumor tissue was detected by immunohistochemistry. The subjects could proceed to the subsequent clinical trial if the NY-ESO-1 immunohistochemistry was positive. Each subject received only one cell reinfusion.

ELIGIBILITY:
Inclusion Criteria:

1. Sign informed consent before conducting any trial-related activities;
2. Age of 18-75 years old, male or female;
3. Patients with first-line treatment failure;
4. Measurable lesions according to RECIST1.1 criteria.
5. During the trial screening period, the following two screening criteria must be met (by the sponsor) :

   * HLA-A*02 positive;
   * The positive rate of NYESO-1 immunohistochemical staining was ≥20%.
6. ECOG score 0-1;
7. The expected survival time is more than 3 months;
8. Antineoplastic drugs and treatments were not allowed for 4 weeks before TCR-T cell infusion;
9. Echocardiography showed left ventricular ejection fraction ≥50%;
10. Laboratory test results should at least meet the following specified indicators:

    * WBC ≥3.0×109/L;
    * Absolute neutrophil count (ANC) ≥1.5×109/L;
    * Absolute lymphocyte count (ALC) ≥1.0×109/L;
    * platelet (PLT) ≥75×109/L;
    * hemoglobin ≥10g/dL (no blood transfusion in the past 7 days);
    * Prothrombin time or INR≤1.5x upper limit of normal unless receiving anticoagulant therapy;
    * Partial prothrombin time (APTT) ≤1.5x upper limit of normal time, unless receiving anticoagulant therapy;
    * 24-hour creatinine clearance ≥60mL/ min;
    * Aspartate aminotransferase (AST/SGOT) ≤2.5×ULN;
    * alanine aminotransferase (ALT/SGPT) ≤2.5×ULN;
    * Total bilirubin (TBIL) ≤1.5×ULN
11. Negative pregnancy tests in women of childbearing potential prior to study treatment; Consent must be given to use effective contraception during treatment.
12. During the whole period of the trial, I can regularly visit the enrolled research institutions for relevant testing, evaluation and management.

Exclusion Criteria:

1. Patients who received major surgery, conventional chemotherapy, large area radiotherapy, immunotherapy or biological therapy within 4 weeks before entering the trial;
2. Known to produce allergic reactions to any component of the trial treatment;
3. no recovery from previous surgery or treatment-related adverse events to ≤ grade 2 CTCAE;
4. Poorly controlled hypertension (systolic blood pressure > 160mmHg and/or diastolic blood pressure > 90mmHg) or clinically significant (e.g., active) cardio-cerebrovascular disease; Cerebrovascular accident (within 6 months before the signing of informed consent), myocardial infarction (within 6 months before the signing of informed consent), unstable angina, congestive heart failure of New York Heart Association class II or higher (Appendix), or severe arrhythmia that could not be controlled with medications or that had the potential to affect study treatment; Electrocardiogram (ECG) was significantly abnormal or the mean QTc interval was ≥450 msec on three consecutive occasions.
5. Combined with other serious organic diseases and mental disorders;
6. Have active systemic infection requiring treatment, including active tuberculosis, known HIV positivity, or clinically active hepatitis A, B, or C; (Virus carriers should be excluded)
7. Patients with autoimmune diseases: those with a history of inflammatory bowel disease or a history of autoimmune diseases (such as systemic lupus erythematosus, vasculitis, and invasive lung disease) judged by the investigators to be not suitable for this study should be excluded; (Patients with vitiligo are not excluded).
8. Administration of chronic systemic cortisone steroids, hydroxyurea, and immunomodulatory agents (e.g., interleukin-2, interferon-α or γ, GM-CSF, mTOR inhibitors, cyclosporine, thymosin, etc.) within 4 weeks prior to cell therapy."
9. History of organ transplantation, autologous/allogeneic stem cell transplantation and renal replacement therapy;
10. Known uncontrolled diabetes mellitus, pulmonary fibrosis, interstitial lung disease, acute lung disease or liver failure;
11. Known alcohol and/or drug abuse;
12. Pregnant or lactating women;
13. Trial participants with any coexisting medical conditions or diseases judged by the investigators to be likely to impair the conduct of the trial;
14. No legal capacity/limited capacity.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-05-22 (Actual); Primary Completion 2027-04-25 (Estimated); Study Completion 2027-06-25 (Estimated)

PRIMARY OUTCOMES:
DLT | Up to 28 Days
  Determining the dose-limiting toxicity (DLT) of Super1 TCR-T adoptive Immunotherapy
MDT | Up to 28 Days
  Determining the maximum Tolerated dose (MTD) of Super1 TCR-T adoptive Immunotherapy

SECONDARY OUTCOMES:
ORR | One year after cell reinfusion
  Objective response rate,defined as the proportion of subjects with a confirmed PR or better best response
OS | One year after cell reinfusion
  overall survival，time from subject's treatment to death. Participants with no death recorded at the time of statistical analysis were censored at the time of the last follow-up. In cases of loss to follow-up, data were censored at the date of the last contact with the participant.
PFS | One year after cell reinfusion
  progression-free survival ，the time from the subject's treatment to the occurrence of PD or death from any cause, whichever occurred first. If no event (PD or death) occurred, the date of the last response assessment was the censored time for PFS.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Gaungdong, China